CLINICAL TRIAL: NCT05414942
Title: Opioid Reduction Program for Total Knee Replacement Patients
Acronym: TKR ORP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: Campbell Clinic (Other)
Responsible Party: Principal Investigator, Karen Derefinko, PhD, Associate Professor, University of Tennessee
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 21-08206-XP
Record Dates: First submitted 2022-06-01; First posted 2022-06-10 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Knee Injuries; Knee Injuries and Disorders; Opioid Use
Keywords: Opioid; Total Knee Replacement; Knee Arthroplasty; Knee Injuries; Prevention; Analgesics, Opioid
MeSH Terms: conditions — Knee Injuries; Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment As Usual (TAU) (No Intervention): No intervention will be administered.
- Opioid Reduction Program (Experimental): Participants will engage in a brief, educational intervention pre-surgery and a brief booster session 2 weeks post-surgery.
  Interventions: Behavioral: Opioid Reduction Program

INTERVENTIONS:
Behavioral: Opioid Reduction Program — Subjects will engage in a brief, educational session which includes information about the appropriate use of opioid pain medication, exposure and tolerance, the definition of misuse and opioid-related harms, how to wean off medication, alternative pain management strategies, and appropriate disposal of leftover medication.
  Other Names: TKR-ORP
  Arms: Opioid Reduction Program

SUMMARY:
In the context of prescribed opioids, research suggests that increased exposure is associated with long-term opioid use. Orthopedic surgeries are associated with the prescribing of more opioid narcotics than any other surgical specialty, particularly for Total Knee Replacement surgery, which is associated with severe post-operative pain. The proposed project is a randomized clinical trial to explore the efficacy of our Total Knee Replacement Opioid Reduction Program (ORP) vs. Treatment As Usual (TAU) in the reduction of opioid use following total knee replacement surgery.

DETAILED DESCRIPTION:
The purpose of the study is to build upon our existing research to: (1) explore the efficacy of a disseminable Opioid Reduction Program (ORP) to reduce long-term use of prescribed opioids following TKR surgery, (2) assess whether lower opioid use following surgery is related to better functional recovery, and (3) model opioid use trajectories following TKR surgery (i.e., MMEs/week for 12 weeks), which will allow us to examine the factors that characterize at-risk groups.

There will be one control arm (Treatment as Usual or TAU) and one experimental arm (Opioid Reduction Program or ORP). The experimental arm will receive the intervention material twice. The first session is pre-surgery, and the second session is a shortened "booster" session approximately 2-weeks post-op.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older.
* Presenting for a total knee replacement (TKR) surgery at Campbell Clinic which will result in an opioid prescription.
* Access to a telephone.
* Able to consent in English.

Exclusion Criteria:

* Under the age of 18.
* Contraindications to use of opioid medication.
* No access to a telephone.
* Unable to understand consent materials in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Opioid pills (dose and type) prescribed by Campbell Clinic. | 12-weeks post-op.
  transcribed from medical record at Campbell Clinic
Opioid pills prescribed outside of Campbell Clinic. | 12-weeks post-op.
  assessed via scan of prescription drug monitoring database for Tennessee
Opioid pill count questionnaire. | 12-weeks post-op.
  self-report from participant of how many opioids are left in the bottle at the 12 week assessment

SECONDARY OUTCOMES:
KOOS Jr. | 12-weeks post-op.
  There are 3 domains scored from the 7-item measure: Stiffness (1 item), assessed on a 1-5 scale from None to Extreme; Pain (4 items), assessed on a 1-5 scale from None to Extreme; Function, daily living (2 items), assessed on a 1-5 scale from None to Extreme

CONTACTS AND LOCATIONS:
Overall Officials: Karen Derefinko, PhD, Principal Investigator — University of Tennessee
Locations (1):
- University of Tennessee Health Science Center, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
It is anticipated that a cleaned data set of study-specific data will be provided within two years following the termination of the study for the data archive and this data set would be made public. Confidentiality of individual participants would be maintained with all releases of data. The final study analytical database would be processed according to HIPAA definitions for public data sharing. Documentation would be provided along with the data sharing file that includes but is not limited to: data dictionary, data codebook, valid variable ranges (where provided), the protocol, procedure and operational manuals, intervention manual or programs and any electronic versions of any paper forms that were used in data collection.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2 years after data collection ends

DOCUMENTS (3):
  • Study Protocol (2021-10-05): https://cdn.clinicaltrials.gov/large-docs/42/NCT05414942/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/42/NCT05414942/SAP_001.pdf
  • Informed Consent Form (2021-06-24): https://cdn.clinicaltrials.gov/large-docs/42/NCT05414942/ICF_002.pdf